CLINICAL TRIAL: NCT06996223
Title: A Multicenter, Prospective, Randomized Controlled Trial to Evaluate the Efficacy of PCSK-9 Inhibitors in Delaying the Progression of Calcified Aortic Valve Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFEC-2025-177
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Aortic Stenosis; PCSK9 Inhibitor; Calcified Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Subjects randomized to the experimental group will be treated with a lipid-lowering regimen based on PCSK9 inhibitors (subcutaneous injection, twice a week) + statins (maximum tolerated dose).
  Subjects randomized to the control group will be treated with a lipid-lowering regimen based on statins (the maximum tolerated dose).
  The study lasted for 4 years, and the patients were followed up at 1, 6, 12, 24, 36, and 48 months to assess the efficacy and safety of the drug administration and to collect information on relevant examinations and tests.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Subjects randomized to the group A will be treated with a lipid-lowering regimen based on PCSK9 inhibitors (subcutaneous injection, twice a week) + statins (maximum tolerated dose).
  The study lasted for 4 years, and the patients were followed up at 1, 6, 12, 24, 36, and 48 months to assess the efficacy and safety of the drug administration and to collect information on relevant examinations and tests.
  Interventions: Drug: The Group A received PCSK9 inhibitor plus statin therapy
- Group B (No Intervention): Subjects randomized to the B group will be treated with a lipid-lowering regimen based on statins (the maximum tolerated dose).
  The study lasted for 4 years, and the patients were followed up at 1, 6, 12, 24, 36, and 48 months to assess the efficacy and safety of the drug administration and to collect information on relevant examinations and tests.

INTERVENTIONS:
Drug: The Group A received PCSK9 inhibitor plus statin therapy — Subjects randomized to the Group A will be treated with a lipid-lowering regimen based on PCSK9 inhibitors (subcutaneous injection, twice a week) + statins (maximum tolerated dose).
  Arms: Group A

SUMMARY:
The aim of this clinical trial is to understand whether the drug PCSK9 inhibitor can slow the progression of calcific aortic valve disease and to understand the safety of the drug.

The primary objective of the study was to evaluate whether PCSK9 inhibitors could delay the progression of aortic stenosis in patients with aortic stenosis.

Secondary objectives: 1) To evaluate whether PCSK9 inhibitors can delay the progression of valve calcification in patients with aortic stenosis;2) To evaluate whether PCSK9 inhibitors can reduce long-term adverse events in patients with aortic stenosis;3) To evaluate the effect of PCSK9 inhibitors on circulating Lp(a) levels in patients with aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign informed consent;
* Age ≥18 years old, gender unlimited;
* Patients with aortic stenosis diagnosed by echocardiography;
* Combined with atherosclerotic cardiovascular disease or
* hypercholesterolemia LDL-C≥4.9mmol/L;
* The blood lipids were not up to standard after the maximum tolerated dose of statins;

Exclusion Criteria:

* Rheumatic aortic stenosis;
* Previous use of PCSK9 inhibitors or allergy to PCSK9 inhibitors;
* Left ventricular ejection fraction ≤35%;
* Patients planned to undergo aortic valve replacement or TAVR in the near future;
* Complicated with other severe valvular diseases;
* Poor adherence to treatment and inability to take medication according to the trial protocol;
* Pregnant and lactating women;
* Combined with active malignant tumors, severe liver and kidney dysfunction and other life expectancy of less than 1 year;
* Participants who are participating in other interventional clinical studies;
* Patients who were judged by the investigator to be ineligible for participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean annual variation of peak aortic valve velocity | Baseline ,6 months,12months,24months,36months,48months,
  Mean annual change in peak aortic valve velocity measured by cardiac ultrasound.

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: SAP, CSR
Time Frame: June 2025 - June 2029